CLINICAL TRIAL: NCT05263050
Title: GU-187: Phase II Trial of Alternative Cabozantinib Dosing Schedule in Metastatic Renal Cell Carcinoma and Neuroendocrine Tumors
Brief Title: Trial of an Alternative Cabozantinib Dosing Schedule in Metastatic Renal Cell Carcinoma and Neuroendocrine Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-1020; GU-187 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Renal Cell Carcinoma; Clear-cell Metastatic Renal Cell Carcinoma; Neuroendocrine Tumors; Carcinoid Tumor
MeSH Terms: conditions — Carcinoma, Renal Cell; Clear-cell metastatic renal cell carcinoma; Neuroendocrine Tumors; Carcinoid Tumor | interventions — cabozantinib; Nivolumab

STUDY DESIGN:
Intervention Model Description: Patients will start at 40 mg of cabozantinib daily and dose escalate or de-escalate based on pre-specified criteria and at set dosing schedules to allow for smaller median dose changes between adjustments.
  Patients in cohorts A and C will be treated with the same cabozantinib alternative dosing schema and schedule, with the exception of Cohort B patients also receiving monthly fix-dosed nivolumab infusions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cabozantinib (Experimental): Cabozantinib treatment will start at 40 mg of cabozantinib daily and dose escalate or de-escalate based on pre-specified criteria and at set dosing schedules to allow for smaller median dose changes between adjustments. The de-escalation would be fine-tuned and adjustments would be made in 10 mg average daily dosing increments by utilizing alternate day dosing schedules (e.g 60 mg/40 mg every other day) rather than decreasing by 20 mg. The maximum dose of cabozantinib is 60 mg daily. Cycles would be 28 days, with weekly follow-up for cycle 1 and bi-weekly follow-up for cycle 2 to allow for prompt dose adjustments, and then monthly. At each check-in, patients that have met the established protocol criteria and were not yet at the maximum dose of 60 mg daily would be eligible for dose-escalation. Patients would also be dose de-escalated as determined by the investigator. Patients who de-escalate may be allowed to re-escalate in the future.
  Interventions: Drug: Cabozantinib
- Cabozantinib and nivolumab (Experimental): Cabozantinib treatment will receive monthly fix-dosed nivolumab infusions, and start at 40 mg of cabozantinib daily and dose escalate or de-escalate based on pre-specified criteria and at set dosing schedules to allow for smaller median dose changes between adjustments. The de-escalation would be fine-tuned and adjustments would be made in 10 mg average daily dosing increments by utilizing alternate day dosing schedules (e.g 60 mg/40 mg every other day) rather than decreasing by 20 mg. The maximum dose of cabozantinib is 60 mg daily. Cycles would be 28 days, with weekly follow-up for cycle 1 and bi-weekly follow-up for cycle 2 to allow for prompt dose adjustments, and then monthly. At each check-in, patients that have met established protocol criteria and were not yet at the maximum dose of 60 mg daily would be eligible for dose-escalation. Patients would also be dose de-escalated as determined by the investigator. Patients who de-escalate may be allowed to re-escalate in the future.
  Interventions: Drug: Cabozantinib; Drug: Nivolumab

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib initiated at 40 mg daily. Dose-escalate or de-escalate based on pre-specified criteria and at set dosing schedules
  Other Names: XL184
Drug: Nivolumab — Nivolumab injection is to be administered as an IV infusion at a dose of 480 mg on day 1 of each cycle
  Other Names: Opdivo
  Arms: Cabozantinib and nivolumab

SUMMARY:
This is a multi-site, three-cohort phase II trial of cabozantinib for IMDC all-risk frontline metastatic renal cell carcinoma (mRCC) patients OR any line mRCC patients who have not previously been treated with cabozantinib, and patients with pancreatic or extra-pancreatic neuroendocrine tumors.

DETAILED DESCRIPTION:
This is a multi-site, three-cohort phase II trial of cabozantinib for IMDC all-risk frontline metastatic renal cell carcinoma (mRCC) patients OR any line mRCC patients who have not previously been treated with cabozantinib, and patients with pancreatic or extra-pancreatic neuroendocrine tumors (NETs). The study is comprised of three cohorts; Cohorts A and C will employ the alternative dosing schema with cabozantinib monotherapy in any-line clear cell or non-clear cell mRCC patients and patients with pancreatic or extra-pancreatic NETs, and Cohort B will employ the alternative dosing schema with cabozantinib in combination with standard-dosed nivolumab in front-line clear cell or non-clear cell mRCC patients.

Study will accrue a total of 111 patients (Cohort A n=49, Cohort B n=37, Cohort C n=25). Patients in cohorts A and C will be treated with the same cabozantinib alternative dosing schema and schedule, with the exception of Cohort B patients also receiving monthly fix-dosed nivolumab infusions. Patients will start at 40 mg of cabozantinib daily and dose escalate or de-escalate based on pre-specified criteria and at set dosing schedules to allow for smaller median dose changes between adjustments. The de-escalation would be fine-tuned and adjustments would be made in 10 mg average daily dosing increments by utilizing alternate day dosing schedules (e.g. 60 mg/40 mg every other day) rather than decreasing by 20 mg (table 1). The maximum dose of cabozantinib is 60 mg daily, while the lowest dosing level on trial will be 20 mg every other day. Cycles would be 28 days, with weekly follow-up for cycle 1 and bi-weekly follow-up for cycle 2 to allow for prompt dose adjustments, and then monthly. At each check-in, patients in Cohorts A and B that have met the established protocol criteria (outlined in Section 6.3) and were not yet at the maximum dose of 60 mg daily would be eligible for dose-escalation. At each check in, patients in cohort C that have met the established protocol criteria and were not yet at the maximum dose of 60 mg daily will be mandated to start next higher dose level. Patients would also be dose de-escalated as determined by the investigator. Patients who de-escalate may be allowed to re-escalate in the future.

ELIGIBILITY:
Inclusion Criteria

* Cohorts A and B: Histologically or cytologically confirmed advanced RCC with any clear cell or non-clear cell component. 100% sarcomatoid is permissible.
* Cohorts A and B: Patient may have had any number of prior therapies for Cohort A, but for Cohort B patients must not have received any systemic therapy in the metastatic setting
* Patients who have received prior (neo)adjuvant immunotherapy with pembrolizumab or similar are eligible for Cohort B IF they completed the adjuvant therapy > 12 months from start of trial therapy
* Treatment naïve patients may be treated in Cohort A if deemed not candidates for nivolumab or if felt single agent cabozantinib most appropriate by the treating clinician
* Cohort C: Well differentiated NET, grades 1-3 (any primary site) who have progressed on or are not eligible for somatostatin analogs per treating physician discretion
* Cohort C: Disease progression within prior 12 months
* Cohort C: Prior or concurrent treatment with somatostatin analogue allowed but no limit on lines of therapy (stable dose of somatostatin for 2 months)

All Cohorts:

* At least one measurable lesion as defined by RECIST version 1.1
* No evidence of pre-existing uncontrolled hypertension as assessed by investigator. Patients may undergo adjustments or additions to their antihypertensive regimen before or during screening to achieve optimal BP control.
* Age > 18 years.
* ECOG performance status 0 - 2
* Patients must have normal organ and marrow function as defined below

  * Leukocytes, > 2,000/mcL
  * Absolute neutrophil count, > 1,500/mcL
  * Platelets, > 100,000/mcL
  * Hgb, > 9 g/dL (>90 g/L)
  * Total bilirubin, ≤ 1.5 x ULN (with the exception of of individuals with Gilberts syndrome who may have a bilirubin <3.0 mg/dL)
  * AST/ALT (SGOT/SGPT)/ALP, < 3 x ULN ALP ≤ 5x ULN with documented bone metastases.
  * Albumin, > 2.8 g/dL
  * Creatinine clearance, > 30 Ml/min/1.73 m2 for patients with creatinine levels above institutional normal
  * PT/INR or PTT, < 1.3 x the laboratory ULN
* Ability to understand and willingness to sign a written informed consent and HIPAA consent document
* Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study treatment

Exclusion Criteria

* Patients who have had systemic anti-cancer therapy or radiotherapy within 14 days or five half-lives, whichever is shorter, prior to entering the study.
* Radiation therapy for bone metastases within 2 weeks, any other radiation therapy within 4 weeks, or systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Ongoing clinically relevant complications from prior radiation therapy would preclude eligibility.
* Patients with prior therapy with cabozantinib.
* Prior systemic therapy directed at advanced RCC is not allowed for patients enrolled to Cohort B (treatment-naïve group).
* Cohort B only: Active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Cohort B only: Patients have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Patients may not be receiving any other investigational agents
* History of allergic reactions or hypersensitivity attributed to compound of similar chemical or biologic composition to the agent(s) used in this study
* Current use or anticipated need for treatment with drugs or foods that are known strong CYP3A4 inhibitors and inducers. Refer to Section 5.3.2 for detailed information. The topical use of these medications (if applicable), such as 2% ketoconazole cream, is allowed.
* Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:
* Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
* Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Cardiovascular disorders:
* Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.
* QTcF > 500 msec within 28 days before first dose of study treatment.
* Uncontrolled hypertension defined as sustained blood pressure (BP) > 160 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment.
* Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before first dose of study treatment.
* Subjects with a diagnosis of incidental, sub-segmental PE or DVT within 6 months are allowed if stable, asymptomatic, and treated with a stable dose of permitted anticoagulation (see exclusion criterion #6) for at least 1 week before first dose of study treatment.
* Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:
* The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.
* Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose of study treatment.

Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment.

* Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.
* Lesions invading or encasing any major blood vessels. Subjects with lesions invading the intrahepatic vasculature, including portal vein, hepatic vein, and hepatic artery, are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Cohort A: Average daily dose of cabozantinib > 42.8 mg in at least 70% of patients | 2 years
  To show that alternative cabozantinib dosing can improve average daily dose compared to historical controls
Cohort B: 75% of patients alive and progression free at 12 months | 1 year
  Cohort B: To show that alternative cabozantinib dosing + nivolumab (standard dose) can improve 12-month rate of progression-free survival over standard dose cabozantinib + nivolumab
Cohort C: Decreased rate of grade ≥ 3 adverse events compared to 75% reported in CABINET trial | 2 years
  Cohort C: To show that alternative cabozantinib dosing can improve rates of grade > 3 adverse events compared to the grade 3-5 adverse events reported in the CABINET trial

SECONDARY OUTCOMES:
Cohort A: Decreased grade ≥ 3 adverse events compared to historical controls (METEOR trial) | 2 years
  Demonstrate that alternative dosing can change overall toxicity compared to historical controls by monitoring grade ≥ 3 adverse events compared to historical controls
Cohort A: Improved median duration of time on drug compared to historical controls | 2 years
  Show that alternative scheduling can change median duration of time on drug compared to historical controls
Cohort A: Objective response rate per RECIST 1.1 criteria of all patients treated | 2 years
  Response rates will be summarized via frequencies and 95% confidence intervals, and compared to historical results using two-sided one-sample exact binomial tests of proportions
Cohort B: Decreased grade ≥ 3 adverse events compared to historical comparison from the CheckMate 9ER trial | 2 years
  Demonstrate that alternative dosing can change overall toxicity compared to historical controls by monitoring grade ≥ 3 adverse events compared to historical controls
Cohort B: Improved median duration on the drug (as defined by time from initiation of therapy to time of cessation of therapy) compared to historical comparison to the CheckMate 9ER trial | 2 years
  Show that alternative scheduling can change median duration of time on drug compared to historical controls
Cohort B: Increased median average daily dose of cabozantinib | 2 years
  Calculate the median average daily dose, and compare it to the null hypothesis using a one-sample Wilcoxon signed-ran test
Cohort B: Objective response rate per RECIST 1.1 criteria of all patients treated | 2 years
  Response rates will be summarized via frequencies and 95% confidence intervals, and compared to historical results using two-sided one-sample exact binomial tests of proportions
Cohort B: Overall Survival analysis of all patients treated within the cohort | 2 years
  Overall survival will be analyzed and summarized using Kaplan-Meier methods and compared to results of historic control using two-sided one-sample log-rank tests
Cohort C: Percent of patients requiring dose reduction as a descriptive endpoint | 2 years
  Percent of patients requiring dose reduction as a descriptive endpoint will be calculated along with the 95% confidence interval.
Cohort C: Progression free survival as a descriptive endpoint | 2 years
  Progression free survival will be characterized as a descriptive endpoint using a Kaplan-Meier curve.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Zibelman, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No